CLINICAL TRIAL: NCT02641847
Title: Efficacy and Safety Study of TA(E)C-GP Versus A(E)C-T for the High Risk Triple-negative Breast Cancer Patients Predicted by the Messenger RNA (mRNA)-Long Non-coding RNA (lncRNA) Signature and Validation of the Signature's Efficacy
Brief Title: TA(E)C-GP Versus A(E)C-T for the High Risk TNBC Patients and Validation of the mRNA-lncRNA Signature
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1506147-4
Record Dates: First submitted 2015-12-22; First posted 2015-12-30 (Estimated); Last update posted 2024-01-25 (Actual); Status verified 2023-09

CONDITIONS: Triple Negative Breast Cancer; Breast Cancer
Keywords: triple negative breast cancer; mRNA-lncRNA signature; chemotherapy; high risk
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Docetaxel; Doxorubicin; Epirubicin; Cyclophosphamide; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High risk group A (Experimental): TA(E)C x 4 cycles to GP x 4 cycles (docetaxel + doxorubicin (epirubicin) + cyclophosphamide to gemcitabine + cisplatin), docetaxel: 75 mg/m2 IV on day 1; doxorubicin: 50 mg/m2 IV on day 1 or epirubicin 75 mg/m2 IV on day 1; cyclophosphamide: 500 mg/m2 IV on day 1; gemcitabine: 1250 mg/m2 IV on day 1 and 8; cisplatin: 75 mg/m2 IV on day 1, dosing interval is 21 days.
  Interventions: Drug: docetaxel; Drug: doxorubicin or epirubicin; Drug: cyclophosphamide; Drug: gemcitabine; Drug: cisplatin
- High risk group B (Active Comparator): A(E)C x 4 cycles to T x 4 cycles (doxorubicin (epirubicin) + cyclophosphamide to docetaxel), doxorubicin: 60 mg/m2 IV on day 1 or epirubicin 90 mg/m2 IV on day 1; cyclophosphamide: 600 mg/m2 IV on day 1; docetaxel: 100 mg/m2 IV on day 1, dosing interval is 21 days.
  Interventions: Drug: docetaxel; Drug: doxorubicin or epirubicin; Drug: cyclophosphamide
- Low risk group C (Other): A(E)C x 4 cycles to T x 4 cycles (doxorubicin (epirubicin) + cyclophosphamide to docetaxel), doxorubicin: 60 mg/m2 IV on day 1 or epirubicin 90 mg/m2 IV on day 1; cyclophosphamide: 600 mg/m2 IV on day 1; docetaxel: 100 mg/m2 IV on day 1, dosing interval is 21 days.
  Interventions: Drug: docetaxel; Drug: doxorubicin or epirubicin; Drug: cyclophosphamide

INTERVENTIONS:
Drug: docetaxel
Drug: doxorubicin or epirubicin
Drug: cyclophosphamide
Drug: gemcitabine
  Arms: High risk group A
Drug: cisplatin
  Arms: High risk group A

SUMMARY:
The purpose of this study is to compare the efficacy and safety between docetaxel combined with doxorubicin (epirubicin) and cyclophosphamide followed by gemcitabine combined with cisplatin and doxorubicin (epirubicin) combined with cyclophosphamide followed by docetaxel for high risk triple negative breast cancer predicted by the mRNA-lncRNA integrated signature and validation the efficacy of the signature.

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) is one of the most aggressive subtypes of breast cancer. Chemotherapy is the current mainstay of treatment. The treatment of patients with TNBC has been challenging due to the heterogeneity of the disease and the absence of well-defined molecular targets. The investigators' previous study has successfully identified and independently validated prognostic and predictive RNA signatures for TNBC, which could be used to classify TNBC patients into high- or low-risk of recurrence. This study is intended to further validate the efficacy of the mRNA-lncRNA signature and also explore better chemotherapy for the predicted high risk TNBC patients.

The current study is designed to validation the efficacy of the mRNA-lncRNA signature and evaluate the efficacy and safety between docetaxel combined with doxorubicin (epirubicin) and cyclophosphamide followed by gemcitabine combined with cisplatin and doxorubicin (epirubicin) combined with cyclophosphamide followed by docetaxel for high risk triple negative breast cancer predicted by the integrated signature.

Primary endpoint for the study: recurrence free survival; second endpoint for the study: safety, disease free survival and overall survival; This open multi-center prospective randomized control study includes TNBC patients with invasive ductal carcinoma. All eligible patients' tumor samples were tested using real-time polymerase chain reaction (PCR) and recurrence risks were predicted using the mRNA-lncRNA signature. Patients with high recurrence risk were randomized to Group A or Group B to receive respective chemotherapy. Among which Group A: TA(E)C x 4 cycles to GP x 4 cycles (docetaxel + doxorubicin (epirubicin) + cyclophosphamide to gemcitabine + cisplatin), docetaxel: 75 mg/m2 IV on day 1; doxorubicin: 50 mg/m2 IV on day 1 or epirubicin 75 mg/m2 IV on day 1; cyclophosphamide: 500 mg/m2 IV on day 1; gemcitabine: 1250 mg/m2 IV on day 1 and 8; cisplatin: 75 mg/m2 IV on day 1, dosing interval is 21 days. Group B: A(E)C x 4 cycles to T x 4 cycles (doxorubicin (epirubicin) + cyclophosphamide to docetaxel), doxorubicin: 60 mg/m2 IV on day 1 or epirubicin 90 mg/m2 IV on day 1; cyclophosphamide: 600 mg/m2 IV on day 1; docetaxel: 100 mg/m2 IV on day 1, dosing interval is 21 days. Patients with low recurrence risk received chemotherapy in Group C: A(E)C x 4 cycles to T x 4 cycles (doxorubicin (epirubicin) + cyclophosphamide to docetaxel), doxorubicin: 60 mg/m2 IV on day 1 or epirubicin 90 mg/m2 IV on day 1; cyclophosphamide: 600 mg/m2 IV on day 1; docetaxel: 100 mg/m2 IV on day 1, dosing interval is 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old
2. Expected survival > 12 months
3. Baseline Eastern Cooperative Oncology Group Performance Status rating 0-1
4. Naïve to chemotherapy or hormonal treatments
5. Pathology confirmed invasive ductal carcinoma of breast
6. Triple negative breast cancer confirmed by pathology
7. No concurrent malignancy (except controlled cervical carcinoma in situ or basal cell carcinoma of skin)
8. No advanced metastasis or metastasis involving brain or liver
9. Adequate bone marrow function, blood routine examination shows neutrophil count ≥ 1.5x109/L, hemoglobin level ≥ 100 g/L, Platelets ≥ 100 x 109/L
10. Adequate liver and kidney function, serum aminotransferase (AST) ≤ 60 Unit/L, serum total bilirubin ≤ 2.5 times Upper Limit of Normal, serum creatinine ≤110μmol/L, urea nitrogen ≤7.1mmol/L
11. No coagulation abnormality
12. Normal heart function, with normal ECG and left ventricular ejection fraction ≥ 55%
13. Women of childbearing age agree to take reliable contraceptive measures during clinical trials, and negative serum or urine pregnancy test within 7 days prior to administration
14. No coagulation abnormality
15. Sign the informed consent statement and voluntarily receive follow-ups, treatments, laboratory tests and other research procedures according to protocol.

Exclusion Criteria:

1. Previous regional or systemic treatment for breast cancer (include but not limited to chemotherapy, radiotherapy, targeted therapy, other clinical trials)
2. Inflammatory breast cancer, bilateral breast cancer or breast cancer already with distant metastasis
3. Complicated with uncontrolled lung disease, severe infection, active peptic ulcer, blood clotting disorders, severe uncontrolled diabetes, connective tissue disorders or bone marrow suppression, and intolerance to neoadjuvant therapy or related treatment
4. Peripheral neuropathy >1 degree caused by any reason
5. History of congestive heart failure, uncontrolled or symptomatic angina, arrhythmias or history of myocardial infarction, refractory hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg);
6. Breast cancer during lactation or pregnancy
7. Mental illness or incompliance to treatment caused by other reasons
8. Known history of severe hypersusceptibility to any agents used in the treatment protocol
9. Patients received major surgery or suffered from severe trauma within 2 months of first administration
10. Currently enroll or recently used (30 days within enrollment) other agent under research or involved in other trial
11. Known to be infected with human immunodeficiency virus (HIV)
12. Other circumstances considered to be inappropriate to be enrolled by researchers

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | three years

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | three years
Recurrence free survival | three years
Overall survival | three years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] He M, Jiang YZ, Gong Y, Fan L, Liu XY, Liu Y, Tang LC, Mo M, Hou YF, Di GH, Liu GY, Yu KD, Wu J, Yan X, Zeng XH, Fu DY, Song CG, Zhuang ZG, Wu KJ, Wang J, Wang ZH, Shao ZM. Intensive chemotherapy versus standard chemotherapy among patients with high risk, operable, triple negative breast cancer based on integrated mRNA-lncRNA signature (BCTOP-T-A01): randomised, multicentre, phase 3 trial. BMJ. 2024 Oct 23;387:e079603. doi: 10.1136/bmj-2024-079603. PMID 39442958